CLINICAL TRIAL: NCT05088291
Title: Effectiveness of a New X-ray Protection Devices in Reducing Radiation in Coronary Intervention Therapy
Brief Title: Application of a New X-ray Protective Device in Coronary Interventional Therapy
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The First People's Hospital of Lianyungang (Other)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 015
Record Dates: First submitted 2021-09-23; First posted 2021-10-21 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Coronary Heart Disease
Keywords: cardiology; coronary angiography; coronary angioplasty; percutaneous coronary intervention; radiation
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The new protection device: A total of 100 patients underwent continuous coronary angiography (CAG) or percutaneous coronary intervention (PCI). The first surgeon does not need to wear a lead dress to stand inside the new protective device (NPD) to perform all operations.
- The traditional lead clothing: A total of 100 patients underwent continuous coronary angiography (CAG) or percutaneous coronary intervention (PCI). The first surgeon wears the traditional lead clothing (TLC) to perform all operations.

SUMMARY:
This is a multi-center, prospective and controlled clinical trial which will enroll 200 coronary arteriography or percutaneous coronary intervention with 2-4 interventional cardiologist. The interventional cardiologist performed 100 interventional procedures using either a new protective device (NPD) or a traditional lead clothing (TLC). The cumulative dose outside the NPD or TLC and the first operator at each height (110cm, 90cm, 50cm, 10cm) was measured. The main indicators of the study are the average X-ray shielding efficiency of the NPD and the TLC at four different heights. The investigators will record all operation information in this study.

DETAILED DESCRIPTION:
In this study, the investigators developed a new protection device (NPD) and compared its effects on the reduction of radiation exposure compared with the traditional lead clothing (TLC).

The NPD (WLXP-006, Yingnuoweite Medical Science and Technology, Co., Ltd., Nanjing, China) is a floor-standing medical radiation protection device mainly composed of a barrel-like frame and protective lead rubber (0.5 mm lead equivalent).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients were admitted to the group for coronary arteriography (CAG) or percutaneous coronary intervention (PCI).

Exclusion Criteria:

* There were no exclusion criteria, and the patients were continuously enrolled for interventional diagnosis and treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for CAG or PCI were successively included in the First Affiliated Hospital of Nanjing Medical University and The First People's Hospital of Lianyungang.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The cumulative absorbed dose at different heights outside the NPD | After study completion, about 6 months
  The 16 thermoluminescent dosimetries (TLD) were placed outside the NPD at a height of 110cm, 90cm, 50cm and 10cm above the ground, with each height divided into four positions (front, back, left and right). After the test, the TLDs were sent to Jiangsu CDC for testing.
The cumulative absorbed dose at different heights outside the TLC | After study completion, about 6 months
  The 12 thermoluminescent dosimetries (TLD) were placed outside the NPD at a height of 110cm, 90cm and 50cm above the ground, with each height divided into four positions (front, back, left and right). After the test, the TLDs were sent to Jiangsu CDC for testing.
The cumulative absorbed dose of the first operator | After study completion, about 6 months
  The 16 thermoluminescent dosimetries (TLD) were placed at a height of 110cm, 90cm, 50cm and 10cm above the ground of the first operator (inside NPD or TLC), and each height is divided into four positions. After the test, the TLDs were sent to Jiangsu CDC for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China